CLINICAL TRIAL: NCT00778427
Title: A Study to Compare the Relative Bioavailability of Ranbaxy and Bristol Myers Squibb Formulations of Metformin 1000 mg Tablets in Healthy Adult Volunteers Under Fasting Conditions
Brief Title: Bioequivalence Study of Metformin Hydrochloride 1000mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy research labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 10640302
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence metformin hydrochloride 1000 mg tablets fasting conditions
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): metformin hydrochloride 1000 mg tablets of Ranbaxy
  Interventions: Drug: metformin hydrochloride 1000 mg tablets
- 2 (Active Comparator): GLUCOPHAGE® (metformin hydrochloride) 1000 mg tablets
  Interventions: Drug: metformin hydrochloride 1000 mg tablets

INTERVENTIONS:
Drug: metformin hydrochloride 1000 mg tablets

SUMMARY:
The objective of this study was to evaluate the relative bioavailability of the test formulation of metformin hydrochloride 1000 mg tablets with an already marketed reference formulation GLUCOPHAGE® (metformin hydrochloride) 1000 mg tablets (Bristol-Myers Squibb Company) under fasted conditions in healthy, male and female adult subjects.

DETAILED DESCRIPTION:
This randomized, single-dose, two-way, crossover study was conducted to compare the relative bioavailability of two formulations of 1000 mg metformin hydrochloride tablets under fasting conditions. The study was conducted with 32 (30 completing) healthy adults in accordance with Protocol No. 10640302 (Revision 0). In each study period, a single dose (1 x 1000 mg tablet) was administered to all subjects following an overnight fast of at least 10 hours. The test formulation was Ohm Laboratories, Inc's (A Group of Ranbaxy Pharmaceuticals Inc.) Metformin Hydrochloride 1000 mg Tablets and the reference formulation was GLUCOPHAGE® (metformin hydrochloride) 1000 mg Tablets (Bristol-Myers Squibb Company). The subjects received the test product in one study period and the reference product in the other period; the order of administration was according to the dosing randomization schedule. There was a 7-day interval between treatments.

Blood samples were collected pre-dose and at intervals over 24 hours after each dose. The plasma samples for all subjects completing both periods of the study were sent to Helen Fassoulas, Director of Operations, Warnex Bioanalytical Services Inc., 3885 boul Industriel, Laval, Quebec, H7L4S3 Canada, Telephone: 450-663-6724, Fax: 450-975-8111 for determination of metformin concentrations.

Statistical analysis was performed by Braulio Suarez, M.D., Novum Pharmaceutical Research Services, Wilcrest Green Office Park, 3320 Walnut Bend Lane, Houston, Texas 77042-4712, USA, Telephone: 832-251-8100, Fax: 832-251-7133.

A total of 32 healthy adult subjects (30 completing).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18 to 60 years of age (inclusive).
2. A body mass index (BMI) of 18-30 kg/m2 inclusive as calculated according to Novum Standard Operating Procedures.
3. Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
4. Signed and dated informed consent form, which meets all criteria of current FDA regulations.
5. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable method of contraception (e.g. condom with spermicide, IUD, hormonal contraceptives) for at least 30 days prior to dosing and during the duration of the study.

Exclusion Criteria:

1. If female, pregnant, lactating or likely to become pregnant during the study.
2. History or allergy or sensitivity to metformin, other hyperglycemic agents, or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
3. Significant history or current evidence of chronic infectious disease, system disorder or organ dysfunction.
4. Presence of gastrointestinal disease or history of malabsorption within the last year.
5. History of psychiatric disorders occurring within the last two years that required hospitalization or medication.
6. Presence of a medical condition requiring regular treatment with prescription drugs.
7. Use of pharmacologic agents known to significantly induce or inhibit drug-metabolizing enzymes within 30 days prior to dosing.
8. Receipt of any drug as part of a research study within 30 days prior to dosing.
9. Drug or alcohol addiction requiring treatment in the past 12 months.
10. Donation or significant loss of whole blood (480 ml or more) within 30 days or plasma within 14 days prior to dosing.
11. Positive test results for HIV, Hepatitis B surface antigen or Hepatitis C antibody.
12. Positive test results for drug of abuse at screening.
13. Positive serum pregnancy test.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-02; Primary Completion 2006-02 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- NovumPharmaceutical Research Services, Las Vegas, Nevada, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html